CLINICAL TRIAL: NCT03269279
Title: Mifepristone and Misoprostol for 2nd Trimester Termination of Pregnancy (13-22 Weeks LMP) in Burkina Faso
Brief Title: Mifepristone and Misoprostol for 2nd Trimester Termination of Pregnancy in Burkina Faso
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1036
Record Dates: First submitted 2017-07-14; First posted 2017-08-31 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Medical; Abortion, Fetus
MeSH Terms: interventions — Mifepristone; Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Medical abortion arm (Experimental): 200mg of Mifepristone and repeat doses of 400mcg of misoprostol every 3 hours administered for medical abortion in 2nd trimester
  Interventions: Drug: Mifepristone; Drug: Misoprostol

INTERVENTIONS:
Drug: Mifepristone — Medication used in conjunction with misoprostol for abortion
  Other Names: Medabon
Drug: Misoprostol — Medication used in conjunction with mifepristone for abortion
  Other Names: Misoclear

SUMMARY:
The goal of this study is to examine the effectiveness and feasibility of a mifepristone-misoprostol medical abortion regimen in terminating pregnancies 13-22 weeks in Burkina Faso.

ELIGIBILITY:
Inclusion Criteria:

* Having an ongoing pregnancy of 13-22 weeks gestation
* Be willing to undergo surgical completion if necessary
* Have no contraindications to study procedures, according to provider
* Be willing and able to consent to participate in the study
* Be willing to follow study procedures
* Respect legal indications for obtaining an abortion

Exclusion Criteria:

* Known allergy to mifepristone or misoprostol/prostaglandin
* Any contraindications to vaginal delivery, including placenta previa
* Previous transmural uterine incsion

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-05-20 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of successful abortion | 24 hours
  Rate of successful abortion, complete evacuation of foetus and placenta with study drugs, within 24 hours of taking misoprostol

CONTACTS AND LOCATIONS:
Overall Officials: Blandine Thieba, MD, Study Director — SOGOB; Evelyne Komboigo, MD, Study Chair — SOGOB
Locations (4):
- Burkina Faso (4):
  - CHUSS, Bobo-Dioulasso
  - CMA Boromo, Boromo
  - CHUYO, Ouagadougou
  - CHR Ouahigouya, Ouahigouya

IPD SHARING:
Plan to Share IPD: No